CLINICAL TRIAL: NCT05694260
Title: An Open-Label Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Bempedoic Acid in Pediatric Patients (6 to 17 Years of Age) With Heterozygous Familial Hypercholesterolemia
Brief Title: A Clinical Study in Children With Heterozygous Familial Hypercholesterolemia (HeFH) Aged 6 to 17 Treated Once Daily With Bempedoic Acid Oral Dosing (CLEAR Path 1)
Acronym: CLEAR Path 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1002-041
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hypercholesterolemia
Keywords: Pediatric; Heterozygous familial hypercholesterolemia; Low-density lipoprotein cholesterol (LDL-cholesterol); Bempedoic acid; ETC-1002; Adenosine triphosphate citrate lyase
MeSH Terms: conditions — Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Participants at 16 to <30 kilograms (kg) body weight at screening receiving once daily 60 milligrams (mg) bempedoic acid for 8 weeks followed by 90 mg bempedoic acid for 8 weeks.
  Interventions: Drug: Bempedoic acid
- Cohort 2 (Experimental): Participants at 30 to 60 kg body weight at screening receiving once daily120 mg bempedoic acid for 8 weeks followed by 150 mg bempedoic acid for 8 weeks.
  Interventions: Drug: Bempedoic acid
- Cohort 3 (Experimental): Participants at greater than 60 kg body weight at screening receiving once daily 180 mg bempedoic acid for 8 weeks.
  Interventions: Drug: Bempedoic acid

INTERVENTIONS:
Drug: Bempedoic acid — Once daily oral dosing with oral tablets.
  Other Names: ETC-1002

SUMMARY:
Multiple-dose study to measure pharmacokinetics, pharmacodynamics and safety of bempedoic acid in pediatric participants 6 to 17 years of age with HeFH.

DETAILED DESCRIPTION:
Dose-selection based on body weight will be determined for use in pediatric clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent(s)/guardian(s) must be willing to provide written informed consent and the participant must provide informed assent before any study-specific procedures are performed;
* Participant must be aged 6-17 years old and willing to swallow tablets;
* Participant must weigh at least 16 kilograms (kg);
* Participant must have a diagnosis of HeFH prior to receiving the first dose of study medication at Treatment Visit T1 per Make Early Diagnosis to Prevent Early Deaths project (MEDPED) criteria by meeting at least one of the following clinical criteria:

  1. Documented diagnosis of HeFH determined by positive genetic testing; or
  2. Documented LDL-C or TC meeting one or more of the following criteria:

  i. LDL-C >200 milligrams per deciliter (mg/dL) (5.2 millimole per liter [mmol/L]) or TC >270 mg/dL (7.0 mmol/L), with no first- second- or third-degree relative with documented FH diagnosis (general population); or ii. LDL-C >155 mg/dL (4.0 mmol/L) or TC >220 mg/dL (5.7 mmol/L), and also having a first-degree relative with documented familial hypercholesterolemia (FH) diagnosis; or iii. LDL-C >165 mg/dL (4.3 mmol/L) or TC >230 mg/dL (5.9 mmol/L), and also having a second-degree relative with documented FH diagnosis; or iv. LDL-C >170 mg/dL (4.4 mmol/L) or TC >240 mg/dL (6.2 mmol/L), and also having a third-degree relative with documented FH diagnosis
* Current treatment with approved stable lipid-modifying therapy (LMT), including an optimal dose of statin with or without other LMT(s), at stable dose for at least 4 weeks prior to Treatment Visit T1 (6 weeks for fibrates; however, gemfibrozil is not allowed in participants taking a statin as per coadministration instructions defined in the statin label). Participants must remain on that stable dose throughout the duration of the trial. Optimal dose of statin will be determined by the investigator using their medical judgment and available sources, including the participant's self-reported history of LMT. A participant's optimal dose of statin is defined as meeting one of the following criteria:

  1. the highest approved dose of statin prescribed for the age of the participant based on regional practice or local guidelines; or
  2. less than the highest approved dose of statin, including no statin, prescribed for the age of the participant based on regional practice or local guidelines (including no statin) if: i. the participant has previously taken 2 or more statin therapies at any dose and not able to tolerate or unresponsive due to their mutations (null); or ii. the participant has previously taken 1 or more statin therapies at any dose and is unwilling to attempt another statin at any dose or advised by a physician to not attempt another statin at any dose.
  3. Participant/parent and investigator attestation to the participant's unwillingness to attempt and/or physician advice to not attempt additional statin therapy will be recorded.

Exclusion Criteria:

* Participant has a diagnosis of homozygous familial hypercholesterolemia (HoFH) or compound HeFH;
* Participant has a fasting triglyceride (TG) level ≥400 mg/dL (4.5 mmol/L);
* Participant has uncontrolled hypothyroidism, including a value for thyroid-stimulating hormone (TSH) < lower limit of normal (LLN) or >1.5 × the upper limit of normal (ULN);
* Participant has liver disease or dysfunction, including:

  1. positive serology for hepatitis B surface antigen (HBsAg) and/or hepatitis C virus antibodies (HCV-AB), or
  2. serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value ≥2 × ULN and/or serum total bilirubin (TB) value ≥2 × ULN. If the serum TB value is ≥1.2 × ULN, a reflex indirect (unconjugated) bilirubin will be obtained and, if consistent with Gilbert's disease or if the participant has a history of Gilbert's disease, the participant may be enrolled in the study.
* Participant has renal dysfunction or glomerulonephritis, including an estimated glomerular filtration rate (eGFR) <75 milliliters/minute/1.73 square meter (mL/min/1.73 m^2).

Other protocol defined inclusion and exclusion criteria.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Plasma trough concentration of ETC-1002 | 8 weeks of steady-state dosing
Area under the plasma concentration-time curve (AUC,ss) of ETC-1002 | 8 weeks of steady-state dosing
Average plasma concentration (Cavg,ss) of ETC-1002 | 8 weeks of steady-state dosing
Maximum plasma concentration (Cmax,ss) of ETC-1002 | 8 weeks of steady-state dosing

SECONDARY OUTCOMES:
Plasma trough concentration of ESP15228 | 8 weeks of steady-state dosing
Plasma concentration at 4 hours (C4hr) of ETC-1002 | Day 1
C4hr of ESP15228 | Day 1
Exposure/LDL-C response relationship | 8 weeks of steady-state dosing
  ETC-1002 dose and exposure/LDL-C-lowering response relationship
Percent change from Baseline in low-density lipoprotein cholesterol (LDL-C) | Baseline and at Weeks 8 and 16
Absolute change from Baseline in LDL-C | Baseline and at Weeks 8 and 16
Percent change from Baseline in non-high-density lipoprotein cholesterol (non-HDL-C) | Baseline and at Weeks 8 and 16
Absolute change from Baseline in non-HDL-C | Baseline and at Weeks 8 and 16
Percent change from Baseline in total cholesterol (TC) | Baseline and at Weeks 8 and 16
Absolute change from Baseline in TC | Baseline and at Weeks 8 and 16
Percent change from Baseline in high-sensitivity C-reactive protein (hsCRP) | Baseline and at Weeks 8 and 16
Absolute change from Baseline in hsCRP | Baseline and at Weeks 8 and 16
Acceptability of taste using a dosing acceptability questionnaire | Up to Week 16
Acceptability of ease of swallowing using a dosing acceptability questionnaire | Up to Week 16
Number of participants reporting Serious adverse events (SAEs) and non-SAEs | Up to Week 16

CONTACTS AND LOCATIONS:
Locations (24):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Providere Research Inc, West Covina, California
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Washington University School of Medicine, Division of Endocrinology, Metabolism and Lipid Research, St Louis, Missouri
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cardiology Care for Children, Lancaster, Pennsylvania
  - University of Utah and Primary Children's Hospital, Salt Lake City, Utah
- Canada (3):
  - University of Alberta Hospital - Stollery Children's Hospital, Edmonton, Alberta
  - McMaster University Medical Center, Hamilton, Ontario
  - Ecogene-21, Chicoutimi, Quebec
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Viborg Regional Hospital, Viborg
- Germany (2):
  - Universitaetsklinikum Frankfurt - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt am Main
  - Kinder- und Jugendkrankenhaus AUF DER BULT, Hanover
- Netherlands (2):
  - Amsterdam UMC - Locatie AMC, Amsterdam
  - Erasmus MC, Rotterdam
- Spain (7):
  - Hospital Abente y Lago, A Coruña, Galicia
  - Corporacio Sanitaria Parc Tauli - Hospital de Sabadell, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario de Jerez de la Frontera, Cadiz
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No
The Investigator must ensure that the participant's confidentiality is maintained. The names and identities of all research participants will be kept in strict confidence and will not appear on eCRFs or other records that are provided to or retained by the Sponsor (or designee). If a participant's name appears on any document, it must be redacted and replaced with the participant identifier before a copy of the document is supplied to the Sponsor (or designee). The ICF must include appropriate statements explaining that participant data will be confidential and the actions that will be taken to ensure participant confidentiality.
  Any other confidentiality requirements specified by the site, IRB or IEC, or national or local regulations will be adhered to and detailed appropriately in the ICF.